CLINICAL TRIAL: NCT01232608
Title: Exercise Training in Patients With Coronary Heart Disease and Type 2 Diabetes
Acronym: EXCADI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/1060-1
Record Dates: First submitted 2010-10-25; First posted 2010-11-02 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus, Type 2; Atherosclerosis
Keywords: Coronary Artery Disease; Atherosclerosis.; Diabetes Mellitus, type 2; Exercise; HbA1c; Carotid Atherosclerotic Disease; Inflammation
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2; Atherosclerosis; Motor Activity; Carotid Artery Diseases; Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): 12 months of exercise training
  Interventions: Behavioral: Exercise
- Control (No Intervention): Normal follow-up by primary physician

INTERVENTIONS:
Behavioral: Exercise — 12 months of exercise training
  Arms: Exercise

SUMMARY:
Diabetes mellitus (DM) is an important risk factor in the development of cardiovascular disease, and people with type 2 diabetes have a two- to four-fold increased risk for cardiovascular morbidity and mortality. Physical activity is a well established therapeutic modality for type 2 diabetes. In patients with coronary artery disease (CAD), several clinical trials have shown reduced mortality and reduced progression of atherosclerosis with lifestyle intervention including physical activity. But few studies have investigated the effect of physical training in patients suffering from both diseases.

The aim of this study is to investigate the effect of one year of organized physical exercise in patients with both coronary heart disease and type 2 diabetes on glucometabolic state and progression of atherosclerosis.

The project is a randomized, controlled, open study on physical exercise. 136 patients will be randomized at inclusion to a physical exercise group or a control group, the latter with "normal" follow-up and not discouraged form physical activity. The intervention period will be 12 months, and the physical training program will be developed and conducted in collaboration with Norwegian School of Sport Sciences. The inclusion of patients started summer 2010, the exercise program begins in September 2010 and the practical issues of the study is planned to end during spring 2012.

The main hypothesis is that physical exercise improves the glucometabolic state and reduces progression of atherosclerosis in patients with coronary heart disease and type 2 diabetes, and secondary that physical exercise induces favourable changes in cardiovascular risk factors, use of medication, and co-morbidity associated with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease
* type 2 diabetes

Exclusion Criteria:

* serious diabetic retinopathy, nephropathy and/ or neuropathy
* other serious diseases like cancer, stroke or MI last three months, unstable angina, decompensated heart failure, serious ventricular arrhythmia, aortic aneurism, serious valvular heart disease, chronic obstructive pulmonary disease GOLD classification IV, deep venous/ pulmonary embolism, ongoing infections, serious musculoskeletal disorders.
* other serious limitations to physical exercise
* pathological exercise stress test warranting further cardiovascular examination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Glucometabolic state | 12 months
  Glucometabolic state is defined as: HbA1c, fasting insulin, fasting c-peptid, fasting blood glucose
Atherosclerosis | 12 months
  Atherosclerosis will be assessed by measurements of:
  * Carotid intima-media thickness (IMT)
  * Biomarkers of inflammation, haemostasis and endothelial function

SECONDARY OUTCOMES:
Dyslipidemia | 12 months
  Dyslipidemia will be measured by total cholesterol, HDL, LDL, fasting triglycerides and free fatty acids
Visceral obesity | 12 months
  Visceral obesity will be measured by waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Ingebjørg Seljeflot, phd professor, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Ullevål, Oslo, Norway

REFERENCES:
- [Derived] Zaidi H, Byrkjeland R, Njerve IU, Akra S, Solheim S, Arnesen H, Seljeflot I, Opstad TB. Adiponectin in relation to exercise and physical performance in patients with type 2 diabetes and coronary artery disease. Adipocyte. 2021 Dec;10(1):612-620. doi: 10.1080/21623945.2021.1996699. PMID 34779349
- [Derived] Aune SK, Byrkjeland R, Solheim S, Arnesen H, Troseid M, Awoyemi A, Seljeflot I, Helseth R. Gut related inflammation and cardiorespiratory fitness in patients with CAD and type 2 diabetes: a sub-study of a randomized controlled trial on exercise training. Diabetol Metab Syndr. 2021 Apr 1;13(1):36. doi: 10.1186/s13098-021-00655-2. PMID 33794977
- [Derived] Zaidi H, Byrkjeland R, Njerve IU, Akra S, Solheim S, Arnesen H, Seljeflot I, Opstad TB. Effects of exercise training on markers of adipose tissue remodeling in patients with coronary artery disease and type 2 diabetes mellitus: sub study of the randomized controlled EXCADI trial. Diabetol Metab Syndr. 2019 Dec 19;11:109. doi: 10.1186/s13098-019-0508-9. eCollection 2019. PMID 31890043